CLINICAL TRIAL: NCT01394458
Title: Efficacy and Safety of an Ethanol/Sodium Citrate Locking Solution to Prevent Hemodialysis Catheter-Related Infections: A Pilot Study
Brief Title: Efficacy and Safety of an Ethanol/Sodium Citrate Locking Solution: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: MED XL Inc (Unknown); Winnipeg Regional Health Authority (Other)
Responsible Party: Principal Investigator, Dr. Lavern M. Vercaigne, Professor, Faculty of Pharmacy, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Al452-0005
Record Dates: First submitted 2011-07-04; First posted 2011-07-14 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2015-12

CONDITIONS: Catheter Related Infection; Bacteremia
Keywords: catheter related infection; bacteremia; hemodialysis
MeSH Terms: conditions — Catheter-Related Infections; Bacteremia | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 30 % ethanol/ 4 % sodium citrate group (Experimental): For patients randomized to the 30% ethanol /4 % sodium citrate group, the lock solution will be provided in pre-filled syringes for single use only. After each dialysis session, the locking solution will be instilled into both catheter lumens, the lumens clamped and caps tightly secured to the hubs. Any remaining 30% ethanol/4% sodium citrate solution in each syringe will be discarded. The locking solution will be withdrawn from the catheter lumens before the next dialysis session.
  Interventions: Other: 30 % ethanol / 4% sodium citrate catheter locking solution
- Heparin 1000 U/ml (Experimental): For patients randomized to the heparin group, the heparin will be provided in 10 ml glass vials. Two, 3 ml syringes will be used to draw up the required volume of heparin to fill each lumen. A separate syringe will be used to fill each catheter lumen. The necessary volume should match the lumen volume with no overfill. The locking solution will be instilled into both catheter lumens, the lumens clamped and caps tightly secured to the hubs. The locking solution will be withdrawn from the catheter lumens before the next dialysis session.
  Interventions: Drug: Heparin 1000 u / ml

INTERVENTIONS:
Other: 30 % ethanol / 4% sodium citrate catheter locking solution — This solution is locked into the lumens of hemodialysis catheters between treatments to prevent infection and thrombosis. Before each dialysis session, the solution should be removed and discarded.
  Other Names: Citra Lok Plus
  Arms: 30 % ethanol/ 4 % sodium citrate group
Drug: Heparin 1000 u / ml — In the control group, heparin 1000 u / ml will be locking into the hemodialysis catheters between treatments to prevent thrombosis. The heparin solution should be removed and discarded before each dialysis session.
  Arms: Heparin 1000 U/ml

SUMMARY:
Currently in Canada, either 4% sodium citrate or heparin 1,000-10,000 U/ml solutions are "locked" into hemodialysis catheters between dialysis sessions to prevent thrombosis. The use of an ethanol/sodium citrate locking solution may have advantages over either of these agents alone. The investigators hypothesize that the 30 % ethanol/4% sodium citrate catheter locking solution is safe and effective in the prevention of catheter-related infections and thrombosis.

DETAILED DESCRIPTION:
The pilot study will utilize a prospective, randomized design. After meeting the inclusion/exclusion criteria and providing written informed consent, patients will be randomly assigned to a 30 % ethanol/ 4% sodium citrate locking solution or heparin 1000 U/ml. Patients will be enrolled from the Health Sciences Centre and the Sherbrook Dialysis Units in Winnipeg, Manitoba, Canada.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Stage V chronic kidney disease preparing to start hemodialysis
* Exchange of an existing catheter to a cuffed, tunneled catheter OR planned vascular access with a cuffed, tunneled catheter
* CVC used for hemodialysis made of alcohol-resistant polymers ie. carbothane

Exclusion Criteria:

* Patients receiving catheters not made of alcohol resistant polymers
* Critically ill patients in ICU setting
* Patients with acute renal failure, who will likely not require prolonged vascular access ( ie. > months)
* Patients with maturing fistulas/graft creation within 2 months
* Patients with planned antibiotic treatment courses lasting longer than 4 weeks from the date of new catheter insertion
* Patients receiving a new cuffed, tunneled catheter over a guide wire, if a fibrin sheath angioplasty was not performed after removing the previous dysfunctional catheter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-08; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Documentation of Serious Adverse Events (SAE) with the use of a 30% ethanol / 4% sodium citrate catheter locking solution. | 6 months
  This outcome will monitor the safety of the ethanol/sodium citrate catheter locking solution.

SECONDARY OUTCOMES:
Rate of catheter-related infections per 1000 catheter days with the 30% ethanol / 4% sodium citrate catheter locking solution compared to heparin. | 6 months
  This outcome will primarily investigate efficacy of the ethanol/sodium citrate locking solution and help to describe effect size for the design of a larger more definitive study.
Rate of catheter dysfunction / 1000 catheter days with the 30% ethanol / 4% sodium citrate catheter locking solution compared to heparin. | 6 months
  Catheter function, defined as blood flow <300 ml/min for 50% of each dialysis session over two consecutive sessions, will be monitored prospectively.
Rate of alteplase use / 1000 catheter days with the 30% ethanol / 4% sodium citrate catheter locking solution compared to heparin. | 6 months
  Need for alteplase use to manage dysfunctional catheters will be documented.

CONTACTS AND LOCATIONS:
Overall Officials: Lavern Vercaigne, Pharm.D., Principal Investigator — University of Manitoba; Lisa Miller, MD, Principal Investigator — University of Manitoba
Locations (1):
- Health Sciences Centre, Winnipeg, Manitoba, Canada

REFERENCES:
- [Derived] Vercaigne LM, Allan DR, Armstrong SW, Zacharias JM, Miller LM. An ethanol/sodium citrate locking solution compared to heparin to prevent hemodialysis catheter-related infections: a randomized pilot study. J Vasc Access. 2016 Jan-Feb;17(1):55-62. doi: 10.5301/jva.5000486. Epub 2015 Dec 7. PMID 26660041